CLINICAL TRIAL: NCT03592836
Title: Diuretic Treatment in High Risk Decompensated Advanced Heart Failure. Bolus Intermittent Versus Continuous Infusion of Furosemide: a Randomized Controlled Trial.
Brief Title: Diuretic Response in Advanced Heart Failure: Bolus Intermittent vs Continuous INfusion
Acronym: DRAIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Simone Frea, MD, Cardiologist, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRAIN trial
Record Dates: First submitted 2018-06-18; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Heart Failure NYHA Class III; Heart Failure NYHA Class IV
MeSH Terms: interventions — Sodium Potassium Chloride Symporter Inhibitors; Furosemide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous infusion of loop diuretics (Active Comparator): Furosemide continuous infusion: 125 or 250 mg die
  Interventions: Drug: Loop Diuretics
- Intermittent infusion of loop diuretics (Active Comparator): Furosemide bolus intermittent: 125 or 250 mg die
  Interventions: Drug: Loop Diuretics

INTERVENTIONS:
Drug: Loop Diuretics — intravenous administration of diuretics
  Other Names: furosemide

SUMMARY:
Loop diuretics are the main therapy for decongestion of patients with advanced acute heart failure. However, these patients often develop diuretic-resistance or even diuretic-refractoriness. In order to overcome such resistance to diuretic, the clinician can increase the dose of furosemide, or change the way of administration (continuous infusion versus boluses) or associate a different class of diuretics (thiazide diuretics, K+-sparing diuretics) up to the addition of low doses of inotropic agents to improve renal perfusion. At the present time there is no evidence in literature in advanced acute heart failure patients about the superiority of the treatment with furosemide in continuous infusion or in intermittent boluses. The aim of the study was to evaluate the efficacy of furosemide in boluses versus continuous infusion in advanced acute heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Advanced heart failure
* WET ≥ 12
* Systolic blood pressure ≤ 110 mmHg
* Serum sodium ≤ 135 mEq/L
* Left systolic ventricular insufficiency (FE < 35%) note for at least 6 months
* Class NYHA III-IV despite medical treatment maximal

Exclusion Criteria:

* Acute coronary syndrome
* Shock cardiogenic
* Chronic renal failure stage V

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Freedom from congestion | 72 hours after randomization

SECONDARY OUTCOMES:
Worsening of renal function | 72 hours after randomization
  Increase in creatinine value > 0.3 mg/dl or increase > 1.5 times
Worsening or persistent HF at 72 h | 72 hours after randomization
  Need to increase the dose of inotropes or diuretics
Change in body weight | 72 hours after randomization
Laboratory data variations in NTproBNP | 72 hours after randomization
Treatment failure | 72 hours after randomization
  Composed by the following events: persistence of congestion, need to increase diuretic treatment, need of renal replacement treatment
Weight differences based on diuretic dose unity | 72 hours after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Simone Frea, MD, Principal Investigator — A.O.U. Città della Salute e della Scienza di Torino
Locations (1):
- Simone Frea, Torino, To, Italy

REFERENCES:
- [Derived] Frea S, Pidello S, Volpe A, Canavosio FG, Galluzzo A, Bovolo V, Camarda A, Golzio PG, D'Ascenzo F, Bergerone S, Rinaldi M, Gaita F. Diuretic treatment in high-risk acute decompensation of advanced chronic heart failure-bolus intermittent vs. continuous infusion of furosemide: a randomized controlled trial. Clin Res Cardiol. 2020 Apr;109(4):417-425. doi: 10.1007/s00392-019-01521-y. Epub 2019 Jun 29. PMID 31256261